CLINICAL TRIAL: NCT04914910
Title: Advanced Hybrid Closed-Loop Treatment in Adults With Type 1 Diabetes Not Meeting Glycaemic Targets: A Randomised Controlled Trial - The Steno 780G Study
Brief Title: The Steno 780G Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Merete Bechmann Christensen, Principal Investigator, MD, PhD, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Steno 780G
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 780G-780G (Experimental): Participants will use MiniMed 780G system for 14 weeks + 14 weeks
  Interventions: Device: Minimed 780G insulin pump
- Usual Care - 780G (Placebo Comparator): Participants will continue with their usual insulin pump for 14 weeks. After completion of the first 14-week periode, they switch to 780G for another 14 weeks.
  Interventions: Device: Minimed 780G insulin pump

INTERVENTIONS:
Device: Minimed 780G insulin pump — This will be a 14-week, open-label, randomised, parallel-group, controlled trial comparing the efficacy of an AHCL system (MiniMed 780G, Medtronic Diabetes, Northridge, CA) with usual care (i.e., a person's usual insulin pump and CGM/isCGM system). After the 14-week trial period, the control group switches to treatment with the MiniMed 780G system. The intervention group continues with the MiniMed 780G system. Both groups are monitored for another 14 weeks.

SUMMARY:
Treatment with insulin pumps and sensor-based glucose monitoring has proven superior to other treatment methods in type 1 diabetes. Still, the majority of people treated with insulin pumps and glucose sensors still does not meet the recommended sensor-based glycaemic targets. Automated insulin delivery systems, also known as closed-loop systems, have shown to improve TIR, TAR, and TBR compared with insulin pump and CGM systems that cannot automatically dose insulin.

The primary objective of the Steno 780G study is to test the effects of the MiniMed 780G system in persons with T1D treated with insulin pump and CGM/isCGM who are not meeting glycaemic targets.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Type 1 diabetes ≥2 years.
* HbA1c >=58 mmol/mol
* Insulin pump treatment ≥12 months
* CGM or isCGM use ≥6 months
* Novorapid use ≥1 week
* Carbohydrate counting and use of the insulin pump bolus calculator for most snacks and meals.
* Carbohydrate intake >80 grams per day (assessed by review of intake recorded in the insulin pump during the 2 weeks prior to the screening visit)

Exclusion Criteria:

* Breast-feeding, pregnancy or planning to become pregnant.
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start.
* Use of hybrid closed-loop systems
* Daily use of paracetamol (acetaminophen)
* Alcohol or drug abuse.
* Severe cardiac disease or retinopathy contraindicating HbA1c <53 mmol/mol.
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the person unsuitable for study participation.
* Lack of compliance with key study procedures at the discretion of the investigator.
* Unacceptable adverse events at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Difference between treatment groups in change in TIR (3.9-10.0 mmol/l) from baseline to Week 14 | From baseline to week 14
  Difference between treatment groups in change in TIR (3.9-10.0 mmol/l) from baseline to Week 14 assessed by 2 weeks of CGM data (12 AM-12 AM (wake + sleep)).

SECONDARY OUTCOMES:
Difference between treatment groups in change in TIR (3.9-10.0 mmol/l) from baseline to Week 14 assessed by 2-week CGM data (6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep)) | From baseline to week 14
Difference in mean glucose | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to Week 14 assessed by 2 weeks of CGM data (each of the endpoints will be calculated for the following 3-time intervals: 6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep), 12 AM - 12AM (wake + sleep)):
Difference in standard deviation | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to Week 14 assessed by 2 weeks of CGM data (each of the endpoints will be calculated for the following 3-time intervals: 6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep), 12 AM - 12AM (wake + sleep)):
Difference in coefficient of variation | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to Week 14 assessed by 2 weeks of CGM data (each of the endpoints will be calculated for the following 3-time intervals: 6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep), 12 AM - 12AM (wake + sleep)):
Percentage of time with glucose values < 3.9 mmol/l (TBR level 1). | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to Week 14 assessed by 2 weeks of CGM data (each of the endpoints will be calculated for the following 3-time intervals: 6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep), 12 AM - 12AM (wake + sleep)):
Percentage of time with glucose values < 3.0 mmol/l (TBR level 2). | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to Week 14 assessed by 2 weeks of CGM data (each of the endpoints will be calculated for the following 3-time intervals: 6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep), 12 AM - 12AM (wake + sleep)):
Percentage of time with glucose values > 10.0 mmol/l (TAR level 1). | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to
Percentage of time with glucose values > 13.9 mmol/l (TAR level 2). | From baseline to week 14
  difference in change in the given variable between treatment groups from baseline to Week 14 assessed by 2 weeks of CGM data (each of the endpoints will be calculated for the following 3-time intervals: 6 AM - 12 AM (wake), and 12 AM - 6 AM (sleep), 12 AM - 12AM (wake + sleep))
Glucose management indicator (an estimate of the laboratory HbA1c value). | From baseline to week 14
  From insulin pump data downloads
HbA1c | From baseline to week 14
Body weight | From baseline to week 14
Total daily insulin dose | From baseline to week 14
  Total daily insulin dose assessed by 2-week insulin pump data downloads
Total daily carbohydrate intake | From baseline to week 14
  Total daily carbohydrate intake assessed by 2-week insulin pump data downloads.

OTHER OUTCOMES:
Number of daily carbohydrate entries in the insulin pump assessed by 2-week insulin pump data downloads | From baseline to week 14
  assessed by 2-week insulin pump data downloads
Hypoglycaemia awareness status. | From baseline to week 14
  Assesed by GOLD and Pedersen-Bjerggaard scale, low scores means aware, high scores means unawareness
Diabetes Treatment Satisfaction Questionnaire scores | From baseline to week 14
  Assessed by Diabetes Treatment Satisfaction Questionnaire. Scores from -36 to 36, high scores means higher satisfaction
Hypoglycaemia Fear Survey scores | From baseline to week 14
  Assessed by Hypoglycemia Fear Survey questionnaire. Scores from 0 to 52, higher scores indicate worse outcome
Diabetes Distress Scale scores | From baseline to week 14
  Assessed by Diabetes Distress Scale questionnaire. DDS consists of 17 items on a 6-point scale. A score of ≥3 indicates a high diabetes distress and a score lower than 3 and ≥2 indicates a moderate diabetes distress.
Pittsburgh Sleep Quality Index scores | From baseline to week 14
  Assessed by PTQI questionnaire
Sleep efficiency (%) assessed by Actigraph GT3x | From baseline to week 14
  assessed by Actigraph GT3x
Physical activity level (sedentary, light, moderate-to-vigorous) assessed by Actigraph GT3x | From baseline to week 14
  assessed by Actigraph GT3x
Difference in number of severe hypoglycaemia events (cognitive impairment requiring external assistance for recovery). | From baseline to week 14
  Assessed by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No